CLINICAL TRIAL: NCT05342779
Title: Radio Frequency Ablation Versus Stripping of Great Saphenous Vein in Management of Primary Varicose Veins , Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Kareem Diaa Eldin AHmed, resident doctor at vascular department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-04-16
Record Dates: First submitted 2022-04-17; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A will undergo stripping of great saphenous vein. . (Active Comparator)
  Interventions: Procedure: stripping of great saphenous vein
- Group B will undergo treatment by radiofrequency ablation. (Active Comparator)
  Interventions: Procedure: stripping of great saphenous vein

INTERVENTIONS:
Procedure: stripping of great saphenous vein — I will make 2 or 3 small cuts in your leg. The cuts are near the top, middle, and bottom of your damaged vein. One is in your groin. The other will be farther down your leg, either in your calf or ankle.
  I will then thread a thin, flexible plastic wire into the vein through your groin and guide the wire through the vein toward the other cut farther down your leg.
  The wire is then tied to the vein and pulled out through the lower cut, which pulls the vein out with it.
  I will close the cuts with stitches. Patient will wear bandages and compression stockings on leg after the procedure.
  Other Names: radiofrequency ablation

SUMMARY:
Varicose veins are one of the most common diseases worldwide it constitutes a progressive disease which during its course it produces complications that usually prompt the patient to seek medical care.

Epidemiological studies of the incidence and prevalence of varicose veins found that the majority of adults would develop it over the course of their lifetime; women were found to be four times likely as men to develop it, the incidence of varicose vein occurrence increases with age.

Varicose veins are defined as tortuous dilated veins after or associated with incompetent valves.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: -. • Adult patients with primary non complicated varicose veins which match the criteria suitable for the procedure

Exclusion Criteria:

* Patients with tortuous GSV that could not allow passage of the sheath, laser fiber, non-palpable distal pulsation.
* inability to ambulate, patients with previous history of deep venous thrombosis (DVT) and pregnant women were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
success rate | one year
  Treatment success was defined as symptomatic improvement as well as decrease in vein diameter,echogenic thickening of vein wall and no flow within the occluded lumen by duplex examination Improvement of symptoms in the treated limb
complication | one year
  * recurrence and recanalization of the treated vein.
  * hyperpigmentation
  * recurrence and recanalization of the treated vein.
  * ecchymosis, paresthesia, hematoma, erythema and phlebitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allegra C, Antignani PL, Bergan JJ, Carpentier PH, Coleridge-Smith P, Cornu-Thenard A, Eklof B, Partsch H, Rabe E, Uhl JF, Widmer MT; International Union of Phlebology Working Group. The "C" of CEAP: suggested definitions and refinements: an International Union of Phlebology conference of experts. J Vasc Surg. 2003 Jan;37(1):129-31. doi: 10.1067/mva.2003.47. No abstract available. PMID 12514589
- [Background] Meissner MH, Gloviczki P, Bergan J, Kistner RL, Morrison N, Pannier F, Pappas PJ, Rabe E, Raju S, Villavicencio JL. Primary chronic venous disorders. J Vasc Surg. 2007 Dec;46 Suppl S:54S-67S. doi: 10.1016/j.jvs.2007.08.038. PMID 18068562
- [Background] Proebstle TM, Vago B, Alm J, Gockeritz O, Lebard C, Pichot O. Treatment of the incompetent great saphenous vein by endovenous radiofrequency powered segmental thermal ablation: first clinical experience. J Vasc Surg. 2008 Jan;47(1):151-156. doi: 10.1016/j.jvs.2007.08.056. PMID 18178468
- [Background] Lurie F, Creton D, Eklof B, Kabnick LS, Kistner RL, Pichot O, Sessa C, Schuller-Petrovic S. Prospective randomised study of endovenous radiofrequency obliteration (closure) versus ligation and vein stripping (EVOLVeS): two-year follow-up. Eur J Vasc Endovasc Surg. 2005 Jan;29(1):67-73. doi: 10.1016/j.ejvs.2004.09.019. PMID 15570274